CLINICAL TRIAL: NCT01147861
Title: A Randomized, Single Blind, Placebo-controlled, Three Period Crossover, Dose Selection Study to Evaluate the Effect of GSK256073, an HM74A Receptor Agonist, on Glucose and NEFA 24 Hour Profile in Type 2 Diabetic Patients.
Brief Title: A Phase 1 Study to Evaluate the Effect of GSK256073, an HM74A Receptor Agonist, on Glucose and NEFA Levels in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 114187
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: T2DM; Pharmacodynamics; GSK256073
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 8-chloro-3-pentyl-1H-purine-2,6(3H,7H)-dione

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Subjects will receive 2 placebo tablets in the morning and 2 placebo tablets in the evening on Day 1 and Day 2.
  Interventions: Other: Placebo
- 5mg BID (Other): Subjects will receive 1 x 5mg tablet and 1 placebo tablet in the morning, and 1 x 5mg tablet and 1 placebo tablet in the evening on Day 1 and Day 2.
  Interventions: Drug: GSK256073
- 10mg QD (Other): Subjects will receive 2 x 5mg tablets in the morning and 2 placebo tablets in the evening on Day 1 and Day 2.
  Interventions: Drug: GSK256073
- 25mg BID (Other): Subjects will receive 1 x 25mg tablet and 1 placebo tablet in the morning, and 1 x 25mg tablet and 1 placebo tablet in the evening on Day 1 and Day 2.
  Interventions: Drug: GSK256073
- 50mg QD (Other): Subjects will receive 2 x 25mg tablets in the morning and 2 placebo tablets in the evening on Day 1 and Day 2.
  Interventions: Drug: GSK256073

INTERVENTIONS:
Drug: GSK256073 — 5mg in the AM and 5mg in the PM
  Arms: 5mg BID
Drug: GSK256073 — 10mg in the AM
  Arms: 10mg QD
Drug: GSK256073 — 50mg in the AM
  Arms: 50mg QD
Drug: GSK256073 — 25mg in the AM and 25mg in the PM
  Arms: 25mg BID
Other: Placebo — 2 placebo tablets in the AM and 2 placebo tablets in the PM
  Arms: Placebo

SUMMARY:
The aim of this study is to verify whether a significant decrease in glucose levels can be achieved with the HM74A agonist GSK256073 in type 2 diabetic patients. Several dose levels and a placebo will be evaluated in a three period crossover study with two active doses and one placebo dose per subject, in order to determine whether there is a dose that produces glucose lowering in the target population. In addition, this study will investigate the optimal dosing regimen for full manifestation of any metabolic effect of GSK256073 by comparing once a day versus twice a day regimens.

DETAILED DESCRIPTION:
This is a multi-center study that will enroll approximately 36 subjects. The study consists of three periods of two days of dosing each. The study will evaluate 5 potential dose regimens. Each subject will receive a randomized sequence of treatments over three periods, with placebo treatment in one period and two different active dose regimens in the other two periods. There will be 5 to 12 days of outpatient washout between treatment periods. Subjects will continue their current treatment on metformin throughout the study. Subjects will monitor blood glucose levels daily via glucometer during oupatient washout periods. A follow-up visit will occur between 5 and 10 days after the last period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented (not less than 6 months prior to screening) type 2 diabetes mellitus diagnosis with:
* HbA1c levels greater than 6.5 percent and less than or equal to 9.5 percent at screening,
* On monotherapy with metformin at the time of screening, and at a todal daily dose greater than or equal to 1000 mg at the time of dosing,
* Fasting plasma glucose level less than 270 mg/dl at screening
* Male or female between 20 and 70 years of age inclusive, at the time of signing the informed consent
* Waist circumference above 102cm (40 inches) for men, and 88cm (35 inches) for women
* Fasting triglycerides between 150 mg/dl and 500 mg/dl, inclusive
* BMI within the range of 22-37 kg/meter squared, inclusive

Exclusion Criteria:

A subject will not eligible for inclusion in this study if any of the following criteria apply:

* Requiring insulin therapy or use of combination oral antidiabetic medications or use of monotherapy other than metformin within the 3 months prior to screening
* Past or present disease (other than type 2 diabetes mellitus) that in the opinion of the Investigator may affect the outcome of this study. These diseases include the following but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, gastrointestinal disease and endocrine disease
* A positive pre-study Hepatitis B surface antigen, or positive Hepatitis C or HIV antibody result within 3 months of screening
* Renal impairment as defined by a calculated GFR less than 60 ml/min
* Any concurrent serious illness (e.g., severe COPD, history of malignancy other than skin cancer within 5 years of initial diagnosis or with evidence of recurrence) that may interfere with a subject completing the study
* Clinical laboratory values as defined per protocol
* ECG parameters as defined per protocol
* History of gout and/or hyperuricemia/uric acid kidney stone or treated with drugs for hyperuricemia: allopurinol and/or probenecid
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Use of the following blood pressure medications or other medications renally excreted via OAT is prohibited: Enalapril (at any dose), Losartan (at any dose), Captopril (at any dose)
* Pregnant females as determined by positive serum hCG test at screening or positive urine hCG test prior to dosing
* Lactating females

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2010-09-07 (Actual); Study Completion 2010-09-07 (Actual)

PRIMARY OUTCOMES:
Weighted mean AUC for glucose | 24 hours

SECONDARY OUTCOMES:
Weighted mean AUC for NEFA, glycerol, triglycerides, insulin, and C-peptide | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Gardens, Florida
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dobbins RL, Shearn SP, Byerly RL, Gao FF, Mahar KM, Napolitano A, Nachbaur GJ, Le Monnier de Gouville AC. GSK256073, a selective agonist of G-protein coupled receptor 109A (GPR109A) reduces serum glucose in subjects with type 2 diabetes mellitus. Diabetes Obes Metab. 2013 Nov;15(11):1013-21. doi: 10.1111/dom.12132. Epub 2013 Jun 12. PMID 23701262
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114187 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114187?search=study&search_terms=114187#rs
- Available data/document: Statistical Analysis Plan: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114187 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register